CLINICAL TRIAL: NCT01279109
Title: Starting Pediatric Obesity Prevention in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00022051
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Pregnancy
Keywords: gestational weight gain
MeSH Terms: conditions — Obesity; Gestational Weight Gain | interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social network building intervention (Experimental): Healthy lifestyle intervention focused on building healthy lifestyle skills and reciprocal social ties between the intervention group members
  Interventions: Behavioral: Social network building intervention
- Home visit (Active Comparator): Home visits focused on preventable infant injuries
  Interventions: Behavioral: Home visit

INTERVENTIONS:
Behavioral: Social network building intervention — Group support and 12 weekly health education/skills building sessions during pregnancy
  Other Names: Madre Sana
  Arms: Social network building intervention
Behavioral: Home visit — Three home visits during pregnancy focused on providing education on infant injury prevention
  Arms: Home visit

SUMMARY:
The purpose of this study is to examine whether we can use social networks to spread health information and health behaviors during pregnancy to prevent excessive gestational weight gain.

DETAILED DESCRIPTION:
The long-term goal of this research is to prevent obesity-related adverse health outcomes for future generations by applying information emerging from social network studies to the development of new population-based behavioral interventions. There are a number of critical periods during fetal development that appear to influence the later development of obesity. Interventions that prevent insult to these critical windows from occurring could improve children's life course trajectories. This project sets the groundwork for examining whether social networks could explicitly be utilized to support women in gaining weight during pregnancy within their clinically recommended weight gain target.

ELIGIBILITY:
Inclusion Criteria:

* any race/ethnicity
* speak Spanish or English
* ≥16 years
* >10 and <28 weeks pregnant
* in prenatal care
* anticipating remaining in Middle Tennessee for their full gestation
* willing to sign a medical information release form so that we can abstract weight measures from their obstetric and pediatric records

Exclusion Criteria:

* speak neither Spanish or English
* <16 years
* < 10 weeks or >28 weeks pregnant
* not in prenatal care
* anticipating leaving Middle Tennessee before full gestation
* unwilling to sign medical information release form
* current or past (within last 12 months) enrollment in another research program that targets weight, physical activity, nutrition

Ages: 16 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabina B Gesell, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Coleman Regional Community Center- Parks & Rec Department, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
An individual participant data set ("The Madre Sana Data Set") and codebook are publically available and can be downloaded at:
  http://www.insna.org/connections/v35/v35_2_6.html Citation: Gesell SB, Tesdahl E. Data Exchange Network: The "Madre Sana" data set. Connections 2016, 35 (2), 62-65.

REFERENCES:
- [Result] Arinze NV, Karp SM, Gesell SB. Evaluating Provider Advice and Women's Beliefs on Total Weight Gain During Pregnancy. J Immigr Minor Health. 2016 Feb;18(1):282-6. doi: 10.1007/s10903-015-0162-8. PMID 25649967
- [Result] Tesdahl E, Gesell SB. Assessing the Impact of De Novo Social Ties within Health Intervention Settings: New Questions for Health Behavior Intervention Research. Clin Transl Sci. 2015 Dec;8(6):676-81. doi: 10.1111/cts.12345. Epub 2015 Nov 18. PMID 26577514
- [Result] Gesell SB, Katula JA, Strickland C, Vitolins MZ. Feasibility and Initial Efficacy Evaluation of a Community-Based Cognitive-Behavioral Lifestyle Intervention to Prevent Excessive Weight Gain During Pregnancy in Latina Women. Matern Child Health J. 2015 Aug;19(8):1842-52. doi: 10.1007/s10995-015-1698-x. PMID 25874878
- [Result] Gesell SB, Tesdahl EA. The "Madre Sana" Data Set. Connect (Tor). 2015;35(2):62-65. doi: 10.17266/35.2.6. No abstract available. PMID 27812234

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 147 were consented; 12 withdrew consent before randomization (reason: too much time to commit); 135 were randomized
Period: Overall Study
Arm/Group | Social Network Building Intervention | Home Visit
Started | 68 | 67
Completed | 55 | 55
Not Completed | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Network Building Intervention | Home Visit | Total
Number analyzed (Participants) | 68 | 67 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (5.9) | 26.3 (5.9) | 26.2 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 67 | 135
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latina | 48 | 50 | 98
  Caucasian | 1 | 5 | 6
  African-American | 15 | 6 | 21
  Asian | 1 | 0 | 1
  Other | 3 | 2 | 5
  Not self-identified | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 68 | 67 | 135
Language preference [Count of Participants; unit: Participants]
  English | 20 | 17 | 37
  Spanish | 41 | 48 | 89
  English AND Spanish | 7 | 2 | 9
Baseline Body Mass Index Category [Number; unit: participants]
  Underweight | 0 | 0 | 0
  Normal weight | 26 | 27 | 53
  Overweight | 23 | 23 | 46
  Obese | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Gestational Weight Gain
Description: Total weight gain during pregnancy extracted from medical record, relative to the 2009 Institute of Medicine (IOM) Weight Gain Recommendations for Pregnancy.
  (Reference: Institute of Medicine (US). Weight gain during pregnancy: reexamining the guidelines. Washington, DC. National Academies Press; 2009. 2009 National Academy of Sciences.)
Time Frame: Duration of pregnancy
Population: Analysis is presented within baseline BMI categories and overall. The Overall Number of Participants Analyzed represents those study participants for whom medical records could be abstracted in the trial (87/135).
Measure: Count of Participants; unit: Participants
Arm/Group | Social Network Building Intervention | Home Visit
Number analyzed (Participants) | 44 | 43
Participants
  Underweight (pre-pregnancy BMI): number analyzed (Participants) | 0 | 0
  Underweight (pre-pregnancy BMI): Under IOM recommendations | 0 | 0
  Underweight (pre-pregnancy BMI): Within IOM recommendations | 0 | 0
  Underweight (pre-pregnancy BMI): Over IOM recommendations | 0 | 0
  Normal weight (pre-pregnancy BMI): number analyzed (Participants) | 15 | 17
  Normal weight (pre-pregnancy BMI): Under IOM recommendations | 8 | 6
  Normal weight (pre-pregnancy BMI): Within IOM recommendations | 6 | 3
  Normal weight (pre-pregnancy BMI): Over IOM recommendations | 1 | 8
  Overweight (pre-pregnancy BMI): number analyzed (Participants) | 14 | 15
  Overweight (pre-pregnancy BMI): Under IOM recommendations | 3 | 6
  Overweight (pre-pregnancy BMI): Within IOM recommendations | 7 | 3
  Overweight (pre-pregnancy BMI): Over IOM recommendations | 4 | 6
  Obese (pre-pregnancy BMI): number analyzed (Participants) | 15 | 11
  Obese (pre-pregnancy BMI): Under IOM recommendations | 4 | 1
  Obese (pre-pregnancy BMI): Within IOM recommendations | 4 | 5
  Obese (pre-pregnancy BMI): Over IOM recommendations | 7 | 5
  All (pre-pregnancy BMI): Under IOM recommendations | 15 | 13
  All (pre-pregnancy BMI): Within IOM recommendations | 17 | 11
  All (pre-pregnancy BMI): Over IOM recommendations | 12 | 19

2. Secondary Outcome: Social Network
Description: Number of discussion partners within the intervention group. Participants were asked to identify by name any program participants with whom they had spoken about their pregnancy or pregnancy-related health behaviors.
Time Frame: 2 times over 12 weeks (Week 6, Week 12)
Population: 59 participants in the intervention group completed at least one wave of social network data collection. Control group participants did not have protocol-specified group sessions to evaluate.
Measure: Mean (Standard Deviation); unit: number of discussion partner ties
Arm/Group | Social Network Building Intervention | Home Visit
Number analyzed (Participants) | 59 | 0
number of discussion partner ties | 3.56 (2.11) |

ADVERSE EVENTS:
Arm/Group | Social Network Building Intervention | Home Visit
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/67
Other Adverse Events (participants affected / at risk) | 0/68 | 0/67

LIMITATIONS AND CAVEATS:
Pilot study; Low session attendance; Missing data from medical record abstractions; Loss to follow-up, possibly due to not requiring participants to attend two baseline visits prior to randomization; Generalizability may be limited to Latina women

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes